CLINICAL TRIAL: NCT05792384
Title: Research on Comprehensive Management of End-stage Severe Chronic Respiratory Diseases - Study of Transbronchial Cryobiopsy in Monitoring Complications of Lung Transplantation
Brief Title: Study of Transbronchial Cryobiopsy in Monitoring Complications of Lung Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ting YANG, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-I2M-1-049-03-TBCB
Record Dates: First submitted 2023-02-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Lung Transplant Rejection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transbronchial cryobiopsy (Experimental): transbronchial cryobiopsy with a 1.1 mm flexible cryoprobe
  Interventions: Procedure: transbronchial lung cryobiopsy with a 1.1 mm flexible cryoprobe
- transbronchial lung biopsy (Active Comparator): transbronchial lung biopsy with biopsy forceps
  Interventions: Procedure: transbronchial lung biopsy with biopsy forceps

INTERVENTIONS:
Procedure: transbronchial lung cryobiopsy with a 1.1 mm flexible cryoprobe — Obtaining lung biopsy samples of patients after lung transplantation through transbronchial lung cryobiopsy with a 1.1 mm flexible cryoprobe
  Arms: transbronchial cryobiopsy
Procedure: transbronchial lung biopsy with biopsy forceps — Obtaining lung biopsy samples of patients after lung transplantation through transbronchial lung biopsy with biopsy forceps
  Arms: transbronchial lung biopsy

SUMMARY:
The goal of this randomized controlled trial is to compare the diagnostic efficacy and safety of transbronchial cryobiopsy (TBCB) and traditional transbronchial lung biopsy for diagnosing the lung transplantation rejection , so as to establish the evidence-based medical basis for the effectiveness and safety of TBCB for monitoring after lung transplantation, It is expected to provide a better auxiliary examination method for lung transplantation.

The main questions it aims to answer are: (1) Histopathological evaluability of specimens; (2) Safety of TBCB; (3) Size and quality of specimen, and number of attempts to obtain five samples.

Participants will undergo TBCB with 1.1 mm flexible cryoprobe or traditional transbronchial lung biopsy with biopsy forceps.

ELIGIBILITY:
Inclusion Criteria:

* Age among 18-65 years old
* After unilateral or bilateral lung transplantation, patient with unexplained pulmonary function decline, acute/chronic clinical lung injury or new pulmonary infiltrates
* or patients requiring monitoring of rejection after lung transplantation
* The patient should undertake routine preoperative examinations for lung cryobiopsy, including routine blood test, coagulation function, electrocardiogram, and chest CT, and the patients have no contraindications to cryobiopsy

Exclusion Criteria:

* patients intolerable to undertake lung biopsy due to severe cardiopulmonary insufficiency or being weak
* The patient is allergic to lidocaine and midazolam
* The patient has recent active massive hemoptysis, or the proposed biopsy site has a high risk of bleeding, such as bronchial artery penetration or suspected renal cancer lung metastasis
* Unstable angina, congestive heart failure, severe bronchial asthma or multiple bullae
* Severe hypertension and arrhythmia, hemodynamic instability and severe respiratory failure (PaO2<60mmHg after oxygen therapy or mechanical ventilation)
* The patient has coagulation disorder and unable to stop taking anticoagulants, antiplatelet drugs, aspirin or non-steroidal anti-inflammatory drugs before lung biopsy
* Suspected aortic aneurysm
* The patient does not agree to participate in this study
* Participating in other studies within three months and not withdrawing or ending
* The researchers think that the patient are not suitable for inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-06 (Estimated); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy of transbronchial cryobiopsy versus traditional transbronchial lung biopsy for diagnosing the lung transplantation rejection | 7 days after lung biopsy
  Diagnostic yield of transbronchial cryobiopsy (TBCB) for diagnosing the lung transplantation rejection, compare with that of traditional transbronchial lung biopsy. The reference standard is the result of Multi-Disciplinary Treatment (MDT).

SECONDARY OUTCOMES:
Incidence of complications | one day, 3 days and 7 days after lung biopsy
  Incidence of complications
Sample size | during surgery
  The area size of the biopsy sample will be measured using the software Image J (version 1.48; Maryland, MD, USA) , and measured in square millimetres.
the number of alveoli in the biopsy sample | 7 days after lung biopsy
  The number of alveoli in the biopsy sample is recorded, according to the histological analysis of the biopsy paraffin section.
the number of blood vessels in the biopsy sample | 7 days after lung biopsy
  The number of blood vessels in the biopsy sample is recorded, according to the histological analysis of the biopsy paraffin section.
the percentage of the area of lung parenchyma without artifacts in the biopsy sample | 7 days after lung biopsy
  The percentage of the area of lung parenchyma without artifacts in the biopsy sample is measured (by the software Image J) and recorded, according to the histological analysis of the biopsy paraffin section.
number of attempts to get five samples | during surgery
  number of attempts to get five samples

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, MD, Principal Investigator — China-Japan Friendship Hospital